CLINICAL TRIAL: NCT06555887
Title: Anterior Discectomy Surgery With Arthrodesis in Degenerative Spinal Canal Stenoses: a Descriptive Pilot Study
Brief Title: Anterior Discectomy Surgery With Arthrodesis in Degenerative Spinal Canal sténoses. (ICASC)
Acronym: ICASC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0183 - ICASC
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Lumbar Canal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single-center retrospective study to characterize changes in the functional capacity of patients (change in Oswestry Desability Index (ODI)) undergoing anterior approach surgery for the management of symptomatic lumbar spinal stenosis between the pre-surgical period and the first assessment 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* anterior surgical management (ALIF or LLIF)
* symptomatic lumbar degenerative pathology (L1-L2 to L5-S1), objectified on MRI (Schizas B, C, D)
* period from June 2017 to December 2019

Exclusion Criteria:

* Traumatic sprains
* History of decompression after the operated stage
* Operated from a later time at the same time
* Scolioses with Cobb angles greater than 10°
* Patients under judicial protection
* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anterior surgery of central lumbar sténoses
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
characterize the evolution of functional capacity in patients undergoing anterior approach surgery for the management of symptomatic lumbar spinal stenosis | 6 month
  Variation in Oswestry Desability Index (ODI) between pre-surgery and first assessment beyond 6 months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three month and ending five years following the end study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.